CLINICAL TRIAL: NCT06320262
Title: Evaluation of the Effect of Wet Cupping (Hijama) on Primary Fibromyalgia Using Brain Magnetic Resonance Spectroscopy and Patient-reported Forms: Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effect of Wet Cupping (Hijama) on Primary Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rasmia Elgohary (Other)
Responsible Party: Sponsor-Investigator, Rasmia Elgohary, assistant professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRC/TDF/01/F
Record Dates: First submitted 2024-02-29; First posted 2024-03-20 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled drugs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): They will receive wet cupping therapy (WCT) every month for 3 consecutive months in addition to a home-based graded exercise program.
  Interventions: Procedure: Wet cupping therapy (WCT)
- Control group (No Intervention): they will receive a home-based graded exercise program, which is comprised of both aerobic and stretching exercises. The patients will be instructed to do the protocols with a gradual increase in both intensity and frequency.

INTERVENTIONS:
Procedure: Wet cupping therapy (WCT) — Type of cupping: Triple-stage wet cupping therapy (Hijama) will be used; sucking, scarification, sucking.
  Cupping points will include one cup on the posterior median line, in the depression below the processus spinosus of the 7th cervical vertebra (Alkahil area); two points in the inter-scapular region 3cm lateral to the lower border of the spinous process of the 3rd thoracic vertebra, two points at inferior angle of the scapula (3cm lateral to lower border of the spinous process of the 7th thoracic vertebra, 2 points at lumbar regions, in addition to the most painful areas.
  After the procedure: Areas of cupping will be covered using sterile gauze. All used tools and materials will be collected in red bags to ensure proper waste disposal. Sharp objects will be disposed of in the sharps disposal box. Telephone follow-up with all patients 48 hours after cupping will be done.
  Other Names: Hijama
  Arms: Intervention group

SUMMARY:
Fibromyalgia has become one of the most prevalent chronic pain conditions that impair quality of life. Wet cupping has gained increasing popularity in treating painful conditions.

This study aims to investigate the effectiveness of wet cupping therapy combined with home-based exercise compared to home-based exercise alone in improving patients diagnosed with primary fibromyalgia syndrome.

DETAILED DESCRIPTION:
Background: The fibromyalgia (FM) syndrome is characterized by widespread chronic pain accompanied by fatigue, cognitive disturbances, sleep disorders, and pronounced somatic and/or psychological distress that impair the quality of life. So far there is no definitive treatment for FM. All available guidelines agreed on the first-line role of non-pharmacological therapies over pharmacological agents.

Cupping therapy (Hijama in Arabic) is an ancient medical art that has been used primarily in the treatment of several painful conditions and has regained popularity in modern medicine.

Purpose: Our study aims to investigate the efficacy of wet cupping therapy in treating patients diagnosed with primary fibromyalgia.

Method: the study will include 50 female patients who had been diagnosed with fibromyalgia syndrome (FMS) according to the American College of Rheumatology (ACR) criteria and had symptoms not exceeding two years.

The eligible patients will further undergo Brain magnetic resonance spectroscopy and clinical assessment including evaluation of the following

1. Widespread pain index (WPI) and pain intensity using a Visual Analog Scale (VAS),
2. Total impact of FM as measured by the validated Arabic version of the Revised Fibromyalgia Impact Questionnaire (FIQR).
3. Evaluation of sleep disturbance using the Jenkins sleep score
4. Evaluation of fatigue using a horizontal line (VAS) anchored by "0=No fatigue " and "100=Worst imaginable fatigue
5. Evaluation of Depression and anxiety using the validated Arabic version of Hospital Anxiety and Depression Scale (HADS)
6. Cognitive function assessment using the Montreal Cognitive Assessment (MoCA)
7. Complete blood count

Randomization: All eligible patients will receive instructions on a home-based graded exercise program, then the patients will randomly be assigned into two groups

1. Control group: will be kept on home-based exercise alone
2. Intervention group: They will receive wet cupping therapy in addition to home-based exercise.

Follow-up assessments: at week 12 after initiating the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-55 years.
* Female individuals to avoid the gender confounding factor.
* Clinical diagnosis of primary fibromyalgia according to the 2016 American College of Rheumatology (ACR) updated diagnostic criteria.
* Moderate pain intensity of ≥ 45 mm or higher on a visual analog scale (VAS).
* No use of skeletal muscle relaxants, antidepressants, antiepileptic drugs, corticosteroids, benzodiazepines, and tramadol within a year before the screening visit.

Exclusion Criteria:

* Underlying rheumatic, malignant, metabolic, hematological, or neurological disorders.
* Patients with bleeding disorders or receiving anticoagulants.
* Previous use, within a year, or current use of skeletal muscle relaxants, antidepressants, antiepileptic drugs, corticosteroids, benzodiazepines, or tramadol
* Patients with BMI ≤ 18 or ≥ 35.
* Pregnant or lactating women.
* Patients with severe anemia.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only female individuals will be included to avoid the gender confounding factor.
Enrollment: 50 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline brain MRS | At the time of inclusion and at week 12
  Voxel placement will be applied to study the following brain centers both thalami, insular regions, amygdalae, hippocampi, superior frontal gyri, and anterior cingulate gyri to determine the concentration of brain neurometabolites Nacetylaspartate (NAA), choline (Cho), and creatine (Cr) and their ratios.

SECONDARY OUTCOMES:
Change from baseline Visual Analog Scale (VAS) | At the time of inclusion and at week 12
  Evaluation of pain using a horizontal line (VAS) anchored by "0=No pain" and "100=Worst pain
Change from baseline in the individual components of the Fibromyalgia Impact Questionnaire Revised (FIQR) | At the time of inclusion and at week 12
  the FIQR is a commonly used instrument in the evaluation of FM patients. It contains 21 questions in 3 domains: function (9 questions), overall impact (2 questions), and symptoms (10 questions), a validated Arabic version will be used.
Change from the baseline sleep disturbance using the Jenkins sleep score (JSS) | At the time of inclusion and at week 12
  Jenkins sleep score (JSS) is a 4-item questionnaire to follow common sleep problems.
  The frequency of sleep problems in the last month is evaluated using four items: difficulty falling asleep, waking up at night, difficulty staying asleep, and non-restorative sleep (ie, waking up after the usual amount of sleep feeling tired and worn out).
  Each item is rated on a Likert-like scale from 0 to 5, where 0 is 'never', 1 is '1-3 days', 2 is 'about 1 night/week', 3 is '2-4 nights/week', 4 is '5-6 nights/week' and 5 is 'almost every night'.
  The total score is a simple sum of all four items' scores and ranges from 0 (no sleep problems) to 20 (most sleep problems). The score of 11 is a cut-off-a score <12 is defined as little sleep disturbances and a score >11 is understood as a high frequency of sleep disturbances.
Change from baseline Fatigue- VAS. | At the time of inclusion and at week 12
  Evaluation of fatigue using a horizontal line (VAS) anchored by "0=No fatigue " and "100=Worst imaginable fatigue
Change from baseline of Hospital Anxiety and Depression Scale (HADS) | At the time of inclusion and at week 12
  The Hospital Anxiety and Depression Scale (HADS) evaluates depression and anxiety, it produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D). Scores greater than or equal to 11 on either scale indicate a definitive case. A validated Arabic version will be used.
Change from baseline of the Montreal Cognitive Assessment (MoCA) | At the time of inclusion and at week 12
  The Montreal Cognitive Assessment score examines seven domains (aspects) of cognitive function (executive/visuospatial function, naming, attention, language, abstraction, recall, and orientation). The maximum score is 30. the score is interpreted as follows; Normal cognition: 26-30 points, Mild cognitive impairment: 18-25 points, Moderate cognitive impairment: 10-17 points, Severe cognitive impairment: Under 10 points.
Change from baseline of the Widespread pain index (WPI) | At the time of inclusion and at week 12
  The widespread pain index evaluates the number of painful areas out of a total of 19 areas, and the number is expected to decrease as the patient improves and vice versa.
Change from baseline hemoglobin | At the time of inclusion and at week 12
  hemoglobin will be assessed in the complete blood count
patient compliance on exercise as instructed | This diary will be reviewed at weeks 4, 8 and 12
  All patients will be asked to complete activity diaries daily to assess adherence. Exercise adherence is considered when the patient can participate in 80% of the prescribed exercise sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Yousef, Professor, Principal Investigator — Kasr Alainy School of Medicine, Cairo University, Egypt; Maha M Sabr, Professor, Principal Investigator — National Research Center (NRC); Dalia B Abdelbaky, A. Prof., Study Chair — National Cancer Institute (NCI); Dalia M Afifi, Consultant, Study Chair — Agouza Rheumatology and Rehabilitation, Armed Forces, Egypt; Gehad G Maghraby, Lecturer, Study Chair — Kasr Alainy School of Medicine, Cairo University, Egypt
Locations (1):
- Rheumatology and Immunology out patient clinic, Internal Medicine Department, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No